CLINICAL TRIAL: NCT00916552
Title: The Effects of Erythropoietin on Depressive Symptoms and Neurocognitive Deficits in Patients With Treatment Resistant Depression and in Patients With Remitted Bipolar Disorder - a Proof of Concept Study
Brief Title: Effects of Erythropoietin on Depressive Symptoms and Neurocognitive Deficits in Depression and Bipolar Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lars Vedel Kessing, professor, MD, DMSc. (Other)
Collaborators: The Ministry of Science, Technology and Innovation, Denmark (Other Government); Novo Nordisk A/S (Industry); University of Oxford (Other); Max-Planck-Institute of Experimental Medicine (Other)
Responsible Party: Sponsor-Investigator, Lars Vedel Kessing, professor, MD, DMSc., Professor, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EPO1
Record Dates: First submitted 2009-06-08; First posted 2009-06-09 (Estimated); Last update posted 2012-11-09 (Estimated); Status verified 2012-11

CONDITIONS: Mood Disorders
Keywords: Erythropoietin; Epo; depression; bipolar disorder; cognition; cognitive function; antidepressant
MeSH Terms: conditions — Mood Disorders; Depression; Bipolar Disorder | interventions — Erythropoietin; Epoetin Alfa; Eosinophil Peroxidase

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Erythropoeitin (Experimental): 40.000 IU, epoetin alfa; Janssen-Cilag
  Interventions: Drug: Erythropoietin

INTERVENTIONS:
Drug: Erythropoietin — 40.000 IU/ml epoetin alfa is administered as intravenous infusions over 15 min weekly for 8 weeks.
  Other Names: Eprex; Epo

SUMMARY:
Depression and bipolar disorder (mania and depression) may be related to problems with nerve cells not being regenerated as fast as normal and are accompanied by cognitive difficulties including memory, attention and planning problems. There is thus a need for better, more efficient treatments with effects on cognitive function. Erythropoietin (Epo) is involved in brain repair and may be a candidate for future treatment strategies. The investigators have demonstrated that a single dose of Epo improves mood and reduces the processing of negative emotional information in healthy volunteers similar to effects seen with antidepressants. With the current study the investigators aim to build upon this discovery by investigating whether repeated Epo administration has antidepressant effects and is able to reverse cognitive difficulties in patients with depression or bipolar disorder. It is hypothesized that Epo will improve mood in treatment-resistant depression and improve cognitive function in this group and in patients with bipolar disorder in remission. If the study reveals beneficial effects of Epo, this would highlight Epo as a candidate compound for future treatment of depression and bipolar disorder, with the potential to directly promote brain repair mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Treatment-resistant depression (defined as failure to respond to at least 2 different types of antidepressants) and an HDRS score of at least 17

OR

* Bipolar disorder in remission (HDRS score of max 14 and Young Mania Scale score of max 14) and subjective complaints of moderate to severe cognitive problems on the Massachusetts General Hospital Cognitive and Physical Functioning Questionnaire (CPFQ) (Fava et al 2006) (score at least 4 on at least 2 domains)
* Unchanged antidepressant or mood stabilizing treatment for at least 2 weeks prior to and during the study

Exclusion Criteria:

* Schizophrenia/ schizoaffective disorder
* Dependence on or abuse of drugs (including alcohol and benzodiazepines corresponding to more than 22.5 mg Oxazepam daily)
* Diabetes
* Renal failure
* Smoking
* Major surgery within 4 weeks prior to inclusion
* Previous Epo-treatment
* Known allergy or antibodies against Epo
* Present or past malignancies
* Epilepsy or epilepsy in first degree family Diagnosis (past or present) of a cardiovascular or cerebrovascular disease
* Untreated or not sufficiently treated arterial hypertension ("therapy-resistant hypertension")
* Initial hematocrit > 50% (males) or > 48% (females)
* Initial platelet count above normal range of laboratory
* Initial reticulocyte count below norma range of laboratory
* Past thromboembolic events or thromboembolic events in first degree family (increased thromboembolic risk)
* Contraindications against prophylactic thrombosis treatment
* Myeloproliferative disorder, polycythemia
* Present immunosuppressive treatment with cyclosporin
* Overweight (BMI > 30) or body weight of less than 45 kg or over 95 kg
* Acute suicidal risk, present or previous suicide attempts in the past 2 years
* Pregnancy or breast feeding
* Women who presently use contraceptive pills
* Sexually active women with child bearing potential who refuse to use double barrier anticonception methods
* Unwillingness or inability to comply with the requirements of the protocol including the presence of any condition (physical, mental, or social) that is likely to affect the subject's ability to comply with the protocol
* Present illness which in investigator's opinion could affect the patient's participation in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2009-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
a) For treatment-resistant depressed patients: Antidepressant effect measured with the Hamilton Depression Rating Scale (HDRS); b) For bipolar patients in remission: Memory measured with the Rey Auditory Verbal Memory Test. | a) Baseline and weeks 5, 9 and 14; b) Baseline and weeks 9 and 14

SECONDARY OUTCOMES:
a) For treatment-resistant depressed patients: number of remissions measured with the HDRS; b) For bipolar patients in remission: sustained attention measured with the RVIP and facial expression recognition. | a) Baseline and weeks 5, 9 and 14; b) Baseline and weeks 9 and 14

CONTACTS AND LOCATIONS:
Overall Officials: Lars V Kessing, Professor, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Copenhagen University Hospital, Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Miskowiak KW, Forman JL, Vinberg M, Siebner HR, Kessing LV, Macoveanu J. Impact of pretreatment interhemispheric hippocampal asymmetry on improvement in verbal learning following erythropoietin treatment in mood disorders: a randomized controlled trial. J Psychiatry Neurosci. 2020 May 1;45(3):198-205. doi: 10.1503/jpn.180205. PMID 31804779
- [Derived] Miskowiak KW, Rush AJ Jr, Gerds TA, Vinberg M, Kessing LV. Targeting Treatments to Improve Cognitive Function in Mood Disorder: Suggestions From Trials Using Erythropoietin. J Clin Psychiatry. 2016 Dec;77(12):e1639-e1646. doi: 10.4088/JCP.15m10480. PMID 27835716
- [Derived] Miskowiak KW, Macoveanu J, Vinberg M, Assentoft E, Randers L, Harmer CJ, Ehrenreich H, Paulson OB, Knudsen GM, Siebner HR, Kessing LV. Effects of erythropoietin on memory-relevant neurocircuitry activity and recall in mood disorders. Acta Psychiatr Scand. 2016 Sep;134(3):249-59. doi: 10.1111/acps.12597. Epub 2016 Jun 3. PMID 27259062
- [Derived] Miskowiak KW, Vinberg M, Glerup L, Paulson OB, Knudsen GM, Ehrenreich H, Harmer CJ, Kessing LV, Siebner HR, Macoveanu J. Neural correlates of improved executive function following erythropoietin treatment in mood disorders. Psychol Med. 2016 Jun;46(8):1679-91. doi: 10.1017/S0033291716000209. Epub 2016 Mar 21. PMID 26996196
- [Derived] Vinberg M, Miskowiak K, Hoejman P, Pedersen M, Kessing LV. The effect of recombinant erythropoietin on plasma brain derived neurotrophic factor levels in patients with affective disorders: a randomised controlled study. PLoS One. 2015 May 26;10(5):e0127629. doi: 10.1371/journal.pone.0127629. eCollection 2015. PMID 26011424
- [Derived] Miskowiak KW, Vinberg M, Macoveanu J, Ehrenreich H, Koster N, Inkster B, Paulson OB, Kessing LV, Skimminge A, Siebner HR. Effects of Erythropoietin on Hippocampal Volume and Memory in Mood Disorders. Biol Psychiatry. 2015 Aug 15;78(4):270-7. doi: 10.1016/j.biopsych.2014.12.013. Epub 2014 Dec 18. PMID 25641635
- [Derived] Miskowiak KW, Ehrenreich H, Christensen EM, Kessing LV, Vinberg M. Recombinant human erythropoietin to target cognitive dysfunction in bipolar disorder: a double-blind, randomized, placebo-controlled phase 2 trial. J Clin Psychiatry. 2014 Dec;75(12):1347-55. doi: 10.4088/JCP.13m08839. PMID 25099079
- [Derived] Miskowiak KW, Vinberg M, Harmer CJ, Ehrenreich H, Knudsen GM, Macoveanu J, Hansen AR, Paulson OB, Siebner HR, Kessing LV. Effects of erythropoietin on depressive symptoms and neurocognitive deficits in depression and bipolar disorder. Trials. 2010 Oct 13;11:97. doi: 10.1186/1745-6215-11-97. PMID 20942940